CLINICAL TRIAL: NCT05761015
Title: A Rehabilitation Walking Program With the Help of a Transient Intake of Nonsteroidal Anti-inflammatory Drug for Patients With Painful Hip/Knee Osteoarthritis - A Pilot Cohort Study With Objectives of Short Walks in the Real Life.
Brief Title: Helping Osteoarthritis Patients to Walk With NSAID
Acronym: PERIPATEI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Plateforme d'Investigation Clinique, INSERM CIC1405, CHU de Clermont-Ferrand, France (Unknown); Fondation Apicil (Other); Médecine Physique et Réadaptation, CHU de Clermont-Ferrand, France (Unknown); Médecine du Sport et Explorations Fonctionnelles, CHU de Clermont-Ferrand, France (Unknown); Rhumatologie, CHU de Clermont-Ferrand, France (Unknown); Direction de la Recherche Clinique et des Innovations, CHU de Clermont-Ferrand, France (Unknown); SARL BOUCHARENC, Saint-Chély d'Apcher, France (Unknown); Inserm U1107 " Neuro-Dol ", Clermont-Ferrand, France (Unknown); Université Clermont-Auvergne, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2022 DUALE
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Chronic Pain
Keywords: Osteoarthritis, Knee; Osteoarthritis, Hip; pain at movement; nonsteroidal anti-inflammatory drug; acetaminophen; paracetamol; personalized medicine; pharmacovigilance
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Chronic Pain

STUDY DESIGN:
Intervention Model Description: cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): there is only one intervention arm and no control arm; the Bayesian analysis will be conducted under hypothetical estimates of superiority vs. control.
  Interventions: Drug: therapeutic program including intermittent drug intake and multimodal rehabilitation program

INTERVENTIONS:
Drug: therapeutic program including intermittent drug intake and multimodal rehabilitation program — The prescribed NSAID molecule shall be chosen according to the patient's risk profile:
  * gastric/duodenal risk: age >65, history of ulcer with remission, history of inflammatory event, current low-dose acetylsalicylic acid treatment ;
  * cardiovascular risk (according to Agostino scale & SCORE);
  The molecule with therefore be:
  * no risk: niflumic acid, 250 mg per intake;
  * gastric/duodenal risk only: diclofenac, 50-100 mg per intake, plus lansoprazole;
  * cardiovascular risk only: ketoprofen, 50-100 mg per intake;
  * double risk: ibuprofen, 200-400 mg per intake, plus lansoprazole. For the walk test, the highest dose of diclofenac or ketoprofen will be used. Then, the patient will be free to half the dose if pain relief is achieved so.
  One gram of acetaminophen will be added to any NSAID intake. The number of intakes will be limited to twice a day (morning and evening) and to 10 times a week.

SUMMARY:
There is a lack of effective analgesic treatments to help walking patients with painful hip/knee osteoarthritis. Our team therefore imagined a new strategy lying on a multimodal rehabilitation walking program with the help of a transient intake of nonsteroidal anti-inflammatory drug (NSAID). NSAIDs are indeed known to act specifically on pain at movement, but their continuous intake would induce unacceptable side effects. To optimize the benefit/risk balance, the molecule to be chosen must fit to the patient's profile, and its intake should cover only the period of interest, i.e. planned walks. Our multimodal rehabilitation program will also include physical techniques such as appropriate footwear, a patient's education aiming at reducing fear/avoidance and spotting side effects of NSAIDs, and a prescription frame to avoid any overdosing.

This clinical study is a single-center, non-randomized, open label, one-arm trial, using drugs prescribed according to their label (i.e. osteoarthritis pain), pending a reinforced monitoring of side effects.

The primary endpoint is to evaluate efficacy and tolerance of a tailored and transient administration of NSAID within a rehabilitation walking program in patients with painful hip/knee osteoarthritis.

Secondary endpoints are to evaluate the adherence to the program and the factors influencing adherence; to identify the less well tolerated conditions of treatment (one condition being one molecule for one patient profile); to identify the factors of success among a set of baseline demographic, morphometric and psychometric variables; and to study the role of central sensitization (assessed by temporal summation) on the efficacy of treatment.

DETAILED DESCRIPTION:
Study schedule:

* Inclusion visit (V0): check of the eligibility criteria, explanation of the protocol, plan for a podiatric consultation, baseline questionnaires, and delivery of diary to collect efficacy outcomes.
* Observation time (4 weeks): baseline measurement of efficacy outcomes (physical activity and pain at walk), podiatric consultation and improvement of footwear (including orthosis or soles).
* Pre-intervention visit (V1) : collection of self-reported outcomes, measurement of temporal summation, 6-min walk test before and after NSAID test *, plan for the first 6-week intervention period and delivery of diary to collect efficacy and tolerance outcomes.
* Intermediate within-intervention visit (after 6 weeks): collection of self-reported outcomes, blood sampling (biological tolerance outcomes), plan for the second 6-week intervention period and delivery of diary to collect efficacy and tolerance outcomes.
* End-of-study visit: collection of self-reported outcomes, blood sampling (biological tolerance outcomes), and collection of last efficacy outcomes (anxiety, depression, kinesiophobia, global impression of change).

  * The patient will undergo two 6-min walk tests at the pre-intervention visit, one before and one 45 min. after oral administration of the NSAID. The patient will be considered as responsive to the NSAID if one of the following criteria occurs: a 15% increase (or more) of the time-to-first pain at walk, self-defined as bothering; a 1-point decrease (or more) of pain intensity (out of 10) throughout the test; or a 15% increase (or more) of the walked distance, if this was < 200 m at the first test. Only patients responsive to the NSAID will continue the trial.

The sequence of successes will be treated in Bayesian analyses. Sequential analyses with be conducted stepwise. At each step, the decision to stop or to keep going will be taken, until a maximum of 50 cases eligible for analysis.

* 1st step (N=20): stop for efficacy if more than 11 successes; stop for non-efficacy if less than 6 successes; continuation otherwise (20 supplementary patients);
* 2nd step (N=40): stop for efficacy if more than 17 successes; stop for non-efficacy if less than 16 successes; continuation otherwise (20 supplementary patients);
* 3rd step (N=50): efficacy if more than 21 successes; non-efficacy otherwise

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral hip or knee idiopathic osteoarthrosis (ACR criteria, Kellgren-Lawrence grade 2 or more on recent X-ray), responsible for pain since 3 at least months, and pain at walking which intensity is at least 4/10 on a numerical rating scale.
* Less than 3 relevant walks (at least 20 minutes or 1000 km) a week.
* Ability to understand and to follow the protocol, and to answer the questionnaires

Exclusion Criteria:

* Pregnancy or breastfeeding
* Legal protection
* Body weight < 40 kg or underweight
* Body weight >120 kg or obesity
* Unability to walk, or unability to walk without support devices (sticks, crutches, orthoses and knee pads are allowed)
* Secondary osteoarthrosis (rheumatism, septic arthritis, recent osteonecrosis, hemochromatosis, gout, acromegalia…).
* Concomitant general bone disease (Paget, Reiter…).
* Concomitant and relevant painful disease else than due to osteoarthrosis (e.g. neuropathic pain, fibromyalgia…)
* Previous recent intervention (e.g. surgery, arthroscopy, joint infiltration) expected to relief osteoarthrosis pain throughout the study period.
* Planned intervention similar to those abovementioned, during the study period.
* Recent initiation of any new analgesic treatment (including systemic steroids).
* Planned initiation of any program expected to relief osteoarthrosis pain during the study period, such as physiotherapy, cognitive behavioral therapy…).
* Planned major surgery during the study period.
* Current cancer disease.
* Immunosuppression.
* Autoimmune disease.
* Concomitant topical or systemic NSAID treatment.
* Chronic strong opioid intake.
* Concomitant insulin therapy.
* Any absolute or relevant contraindication to NSAIDs or acetaminophen, according to the French drug agency

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Success | V1 (pre-intervention visit) + 12 weeks
  success of the therapeutic program (defined by a 30%-increase (or more) of the monthly number of target moves from the baseline observation values, with no treatment discontinuation for NSAID side effects)

SECONDARY OUTCOMES:
Self-declared physical activity (efficacy outcome) | V1 (pre-intervention visit)
  Global Physical Activity Questionnaire (GPAQ)
Self-declared physical activity (efficacy outcome) | V1 (pre-intervention visit) + 6 weeks
  Global Physical Activity Questionnaire (GPAQ)
Self-declared physical activity (efficacy outcome) | V1 (pre-intervention visit) + 12 weeks
  Global Physical Activity Questionnaire (GPAQ)
Actual physical activity (efficacy outcome) | V1 (pre-intervention visit)
  Number of steps per day assessed by pedometer
Actual physical activity (efficacy outcome) | V1 (pre-intervention visit)+ 6 weeks
  Number of steps per day assessed by pedometer
Actual physical activity (efficacy outcome) | V1 (pre-intervention visit) + 12 weeks
  Number of steps per day assessed by pedometer
Pain at walk during the two last weeks (efficacy outcome) | V1 (pre-intervention visit)
  Visual Analogic Scale VAS (11-point numerical rating scale (from 0 = "no pain" to 10) "the worst pain imaginable")
Pain at walk during the two last weeks (efficacy outcome) | V1 (pre-intervention visit) + 6 weeks
  Visual Analogic Scale VAS (11-point numerical rating scale (from 0 = "no pain" to 10) "the worst pain imaginable")
Pain at walk during the two last weeks (efficacy outcome) | V1 (pre-intervention visit)+ 12 weeks
  Visual Analogic Scale VAS (11-point numerical rating scale (from 0 = "no pain" to 10) "the worst pain imaginable")
Patient's Global Impression of Change (efficacy outcome) | V1 (pre-intervention visit) + 12 weeks
  7-item scale
kinesiophobia (efficacy outcome) | V1 (pre-intervention visit) + 12 weeks
  Tampa Scale of Kinesiophobia (TSK)
level of anxious state (efficacy outcome) | V1 (pre-intervention visit) + 12 weeks
  Hospital Anxiety and Depression scale (HADS)
level of depressive state (efficacy outcome) | V1 (pre-intervention visit)+ 12 weeks
  Hospital Anxiety and Depression scale (HADS)

OTHER OUTCOMES:
impairment of renal function (tolerance outcome) | V0 (inclusion)
  either a 15%-increase (or more) of creatininemia from baseline, or a glomerular filtration rate <60 mL.min-1 (MDRD), or creatininemia exceeding 1.5-times the upper limit of the lab's normative values
impairment of renal function (tolerance outcome) | V1 (pre-intervention visit) + 6 weeks
  either a 15%-increase (or more) of creatininemia from baseline, or a glomerular filtration rate <60 mL.min-1 (MDRD), or creatininemia exceeding 1.5-times the upper limit of the lab's normative values
impairment of renal function (tolerance outcome) | V1 (pre-intervention visit)+ 12 weeks
  either a 15%-increase (or more) of creatininemia from baseline, or a glomerular filtration rate <60 mL.min-1 (MDRD), or creatininemia exceeding 1.5-times the upper limit of the lab's normative values
impairment of liver function (tolerance outcome) | V0 (inclusion)
  blood transaminase levels exceeding 2.5-times the upper limit of the lab's normative values, or the occurrence of any relevant abnormality on the liver blood parameters
impairment of liver function (tolerance outcome) | V1 (pre-intervention visit) + 6 weeks
  blood transaminase levels exceeding 2.5-times the upper limit of the lab's normative values, or the occurrence of any relevant abnormality on the liver blood parameters
impairment of liver function (tolerance outcome) | V1 (pre-intervention visit) + 12 weeks
  blood transaminase levels exceeding 2.5-times the upper limit of the lab's normative values, or the occurrence of any relevant abnormality on the liver blood parameters
search for anemia (tolerance outcome) | V0 (inclusion)
  15%-decrease (or more) of hemoglobinemia from baseline
search for anemia (tolerance outcome) | V1 (pre-intervention visit) + 6 weeks
  15%-decrease (or more) of hemoglobinemia from baseline
search for anemia (tolerance outcome) | V1 (pre-intervention visit) + 12 weeks
  15%-decrease (or more) of hemoglobinemia from baseline
relevant digestive event (tolerance outcome) | V1 (pre-intervention visit) + 6 weeks
  persistent gastralgia despite proton-pump inhibitor treatment, or any symptom of hematemesis or rectal bleeding
relevant digestive event (tolerance outcome) | V1 (pre-intervention visit) + 12 weeks
  persistent gastralgia despite proton-pump inhibitor treatment, or any symptom of hematemesis or rectal bleeding
bleeding event (tolerance outcome) | V1 (pre-intervention visit) + 6 weeks
  any abnormal bleeding event if the prescribed NSAID (Non-steroidal anti-inflammatory drugs) is COX (Cyclo-OXygenase inhibitors)-1 selective
bleeding event (tolerance outcome) | V1 (pre-intervention visit) + 12 weeks
  any abnormal bleeding event if the prescribed NSAID (Non-steroidal anti-inflammatory drugs) is COX (Cyclo-OXygenase inhibitors)-1 selective
thrombotic event (tolerance outcome) | V1 (pre-intervention visit) + 6 weeks
  any thrombotic event if the prescribed NSAID is COX-2 selective
thrombotic event (tolerance outcome) | V1 (pre-intervention visit) + 12 weeks
  any thrombotic event if the prescribed NSAID is COX-2 selective
serious adverse event (SAE) (tolerance outcome) | V1 (pre-intervention visit) + 6 weeks
  any SAE considered as relevant by the principal investigator, and possibly due to the intervention
serious adverse event (SAE) (tolerance outcome) | V1 (pre-intervention visit) + 12 weeks
  any SAE considered as relevant by the principal investigator, and possibly due to the intervention
EPICES scale (Evaluation of Precariousness and Health Inequalities in Health Examination Centers) (tolerance outcome) | V0 (inclusion)
  social precarity
Pain Catastrophizing Scale (PCS) (tolerance outcome) | V0 (inclusion)
  pain catastrophizing
Tampa Scale of Kinesiophobia (TSK) (tolerance outcome) | V0 (inclusion)
  kinesiophobia
level of anxious state (tolerance outcome) | V0 (inclusion)
  Hospital Anxiety and Depression scale (HADS)
level of depressive state (tolerance outcome) | V0 (inclusion)
  Hospital Anxiety and Depression scale (HADS)
temporal summation of pain (tolerance outcome) | V0 (inclusion ) + 4 weeks
  measurement both at the forearm ipsilateral to the most painful joint and at the skin area referred to the most painful joint; temporal summation is measured by repeated stimuli with a von Frey filament (180g).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clemront-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No